CLINICAL TRIAL: NCT03512106
Title: The Efficacy of the Acupuncture in the Treatment of Systemic Arterial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: silvia goldmeier (Other)
Responsible Party: Sponsor-Investigator, silvia goldmeier, PhD, Instituto de Cardiologia do Rio Grande do Sul
Organization: Instituto de Cardiologia do Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acupuncture
Record Dates: First submitted 2018-04-10; First posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Arterial Hypertension
Keywords: Arterial Hypertension; Acupuncture
MeSH Terms: conditions — Hypertension | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Chinese traditional acupuncture will be applied.
Who Masked: Outcomes Assessor
Masking Description: Acupuncture sham will be applied (placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Chinese traditional acupuncture
  Interventions: Other: Acupuncture
- Sham group (Placebo Comparator): Sham
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Chinese traditional acupuncture

SUMMARY:
There are few studies in the treatment of hypertension employing acupuncture as a blood pressure regulating technique. The Ministry of Health synthesized the inclusion of integrative and complementary practices within the Unique Health System, such as acupuncture. Our objective is to verify the effect of the acupuncture session on hypertensive patients, measured through ambulatory blood pressure monitoring (ABPM). In this way two groups of patients will be selected in a randomized clinical trial. In the first group, Chinese traditional acupuncture will be applied and in the second group the acupuncture sham will be applied.

DETAILED DESCRIPTION:
Acupuncture as therapy is the subject of conflicting opinions on its effectiveness in scientific means, because in spite of its long existence as a therapeutic tool, raises doubts on the standards of Western science model. In addition, there are few studies in the treatment of hypertension employing Acupuncture as a blood pressure regulating technique. The Ministry of Health synthesized the inclusion of integrative and complementary practices within the Unique Health System, such as Acupuncture. The World Health Organization (WHO) recognizes its effectiveness, having its own concept in the energy imbalance that alter the organic, mental and emotional part addressing a current issue proposing to groundbreaking research. The objective is to verify the effect of the acupuncture session on hypertensive patients, measured through ambulatory blood pressure monitoring (ABPM). In this way two groups of patients will be selected in a randomized clinical trial. In the first group, Chinese traditional acupuncture will be applied and in the second group the acupuncture sham will be applied.

ELIGIBILITY:
Inclusion Criteria:

* patients enrolled in stage I to III of systemic arterial hypertension
* signing the free and informed consent term

Exclusion Criteria:

* patients who do not agree to participate in the study
* patients with systolic pressure values greater than 180 mmHg or diastolic pressure above 110 mmHg
* patients with important comorbidities

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring | 24 hours
  Ambulatory blood pressure monitoring (ABPM) is a feature that enables direct and indirect direct reference to blood pressure in the period 24 or more successive hours with a low level of discomfort throughout the daily activities of the investigated. The possibility of obtaining a representative curve of pressure variations in a given period gives an efficient view of the tension behavior and not simply a static analysis, reflecting only the moment when blood pressure was measured.

IPD SHARING:
Plan to Share IPD: No